CLINICAL TRIAL: NCT03740958
Title: Argatroban Plus R-tPA for Acute Ischemic Stroke: a Prospective, Random, Open Label, Blinded Assessment of Outcome Multi-center Study
Brief Title: Argatroban Plus R-tPA for Acute Ischemic Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Department Chairman, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: k （2018）45
Record Dates: First submitted 2018-11-12; First posted 2018-11-14 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — argatroban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Argatroban combined with rt-PA (Experimental): Drug: Argatroban combined with rt-PA Argatroban as a 100 ug/kg bolus over 3 to 5 minutes was administered intravenously within 1 hour of the tPA bolus followed by a continuous Argatroban infusion of 1.0 ug/kg per minute for 48 hours adjusted to a target activated partial thromboplastin time of 1.75 X baseline (about 10%)
  Interventions: Drug: rt-PA; Drug: Argatroban
- rt-PA (Active Comparator): Drug: rt-PA Intravenous throbolysis with 0.9mg/kg rtPA.
  Interventions: Drug: rt-PA

INTERVENTIONS:
Drug: rt-PA — Intravenous throbolysis with 0.9mg/kg rtPA
Drug: Argatroban — 100 ug/kg bolus over 3 to 5 minutes was administered intravenously, followed by a continuous Argatroban infusion of 1.0 ug/kg per minute for 48 hours adjusted to a target activated partial thromboplastin time of 1.75 X baseline (about 10%)
  Arms: Argatroban combined with rt-PA

SUMMARY:
Acute ischemic stroke (AIS) is the most common type of stroke, which has high rate of morbidity, mortality and disability. A large number of studies have confirmed that the thrombolytic therapy can effectively open blood vessels and improve the functional prognosis of acute ischemic stroke. Therefore, all guidelines recommend intravenous thrombolysis as the first treatment of ischemic stroke patients within 4.5 hours of onset. However, about 1/3 patients receiving thrombolysis will have good prognosis, while a large number of patients will still be disabled and even dead. How to improve the neurological prognosis of thrombolytic patients has been a hot topic in the world.

Recent studies have found that the combined application of argatroban and rt-PA in the treatment of AIS might improve the clinical prognosis and not significantly increase bleeding. Some studies have reported that the combined application of argatroban and rt-PA could improve the blood vessel opening rate, and prevent re-occlusion after opening.

Based on the discussion, the present study is designed to explore the efficacy and safety of argatroban plus rt-PA in the treatment of AIS.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old;
2. Time from onset to treatment ≤4.5 hours;
3. NIHSS ≥ 6
4. Diagnosis of ischemic stroke
5. Signed informed consent by patient self or legally authorized representatives.

Exclusion Criteria:

1. mRS≥2;
2. History of stroke within 3 months;
3. History of intracranial hemorrhage;
4. Suspected subarachnoid hemorrhage;
5. Intracranial tumour, vascular malformation or arterial aneurysm;
6. Major surgery within 1 month;
7. Systolic pressure ≥180 mmHg or diastolic pressure ≥110 mmHg;
8. Platelet count < 105/mm3;
9. Heparin therapy or oral anticoagulation therapy within 48 hours;
10. Abnormal APTT;
11. Thrombin or Xa factor inhibitor;
12. Severe disease with a life expectancy of less than 3 months;
13. Blood glucose < 50 mg/dL (2.7mmol/L);
14. Patients who have received any other investigational drug or device within 3 months;
15. Pregnancy;
16. Researchers consider patients inappropriate to participate in the registry.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 808 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Proportion of mRS (0-1） | 90±7 days

SECONDARY OUTCOMES:
Proportion of mRS (0-2） | 90±7 days
proportion of more than 2 decrease in NIHSS score | 48 hours
  NIHSS, National Institute of Health stroke scale
proportion of early neurological deterioration | 48 hours
  Early neurological deterioration, defined as more than 4 increase in National Institute of Health stroke scale score
Vascular Events | 90±7 days
  The occurence of stroke or other vascular events
symptomatic intracranial hemorrhage | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Huisheng Chen, Doctor, Study Chair — Neurology Department
Locations (1):
- General Hospital of ShenYang Military Region, Shenyang, China

REFERENCES:
- [Derived] Cui Y, Wang EQ, Wang YH, Chen HS. Efficacy of argatroban plus alteplase according to time from onset to thrombolysis in acute ischemic stroke: a prespecified post-hoc analysis of the ARAIS trial. Front Neurol. 2025 Jun 25;16:1582513. doi: 10.3389/fneur.2025.1582513. eCollection 2025. PMID 40635702
- [Derived] Chen HS, Cui Y, Zhou ZH, Dai YJ, Li GH, Peng ZL, Zhang Y, Liu XD, Yuan ZM, Jiang CH, Yang QC, Duan YJ, Ma GB, Zhao LW, Wang RX, Sun YL, Shen L, Wang EQ, Wang LH, Feng YF, Wang FY, Zou RL, Yang HP, Wang K, Wang DL, Wang YL; ARAIS Investigators. Effect of Argatroban Plus Intravenous Alteplase vs Intravenous Alteplase Alone on Neurologic Function in Patients With Acute Ischemic Stroke: The ARAIS Randomized Clinical Trial. JAMA. 2023 Feb 28;329(8):640-650. doi: 10.1001/jama.2023.0550. PMID 36757755
- [Derived] Yang Y, Zhou Z, Pan Y, Chen H, Wang Y; ARAIS Protocol Steering Group. Randomized trial of argatroban plus recombinant tissue-type plasminogen activator for acute ischemic stroke (ARAIS): Rationale and design. Am Heart J. 2020 Jul;225:38-43. doi: 10.1016/j.ahj.2020.04.003. Epub 2020 Apr 8. PMID 32485328